CLINICAL TRIAL: NCT06484946
Title: Pediatric Aquatic Occupational Therapy for Children With Sensory Processing Challenges
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristen Pataki (Other)
Responsible Party: Sponsor-Investigator, Kristen Pataki, Clinical Associate Professor, Cleveland State University
Organization: Cleveland State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Cleveland SU
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Sensory Processing Disorder; Autism Spectrum Disorder; ADHD
Keywords: aquatic therapy; children; sensory processing challenges; aquatics; water; learn to swim; aquatic occupational therapy; occupational therapy; sensory processing
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity | interventions — Occupational Therapy; Aquatic Therapy

STUDY DESIGN:
Intervention Model Description: Every participant receives the intervention. Each child participates in the 8-week aquatic group.
Masking Description: Every participant participated in the aquatic group so the participant, care provider, and investigator were all aware of the intervention provided--therapy in the water.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Aquatic occupational therapy (Experimental): Each child participated and experienced occupational therapy in the water.
  Interventions: Other: aquatic occupational therapy

INTERVENTIONS:
Other: aquatic occupational therapy — Each week, the children participated in a 45-minute aquatic occupational therapy group that consisted of warmup on land, 30 mins of sensory activities in the water, and 10 mins of social activity in the water
  Other Names: occupational therapy; aquatic therapy; social participation

SUMMARY:
Children with sensory processing challenges participated in an 8-week play-based aquatic program addressing goals on behavior, sensory, and participation. It is expected that after the 8-week group, the child's goals will improve demonstrating an effective intervention to address sensory difficulties.

DETAILED DESCRIPTION:
This study examined the effectiveness of an aquatic OT program for children with sensory processing difficulties to develop water readiness skills and improve sensory, behavior, and engagement goals. Six groups of children with deficits in various sensory systems participated in an 8-week aquatic group led by an occupational therapist and occupational therapy students. Each week consisted of a 45-minute aquatic group with a 5 min warmup on land, 30 mins of aquatic activities addressing the sensory system of the week, and 10 mins addressing a social activity with peers. Goals were developed and assessed via the Goal Attainment Scale (GAS). Parents of the participants were given the Sensory Processing Measure (SPM-2) before beginning. As a result of participating in the aquatic OT intervention, percentage of goals achieved will be analyzed. It is expected that this program proves to be beneficial and therefore aquatic OT shows potential for improving sensory processing skills, behavior, and social participation with peers.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ages 4-9 years old
* have an identified sensory processing problem as related on the SPM assessment
* able to maintain head, neck, and trunk control
* able to follow 1-2 step directions

Exclusion Criteria:

* Participants younger than 4 years old and older than 9 years old
* requires lift to get in the water
* difficulty with following 1-step directions

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2024-04-09 (Actual); Study Completion 2024-04-09 (Actual)

PRIMARY OUTCOMES:
Goal Attainment Scaling (GAS) | Scores were tracked weekly for 8 weeks of each program.
  Goals were written on behavior, engagement/participation, and sensory on a scale from -2 (worse outcome) to +2 (better outcome). Each week scores on each goal were documented.
Parent Surveys | Parents were given a post-survey at the 8th week.
  Survey with quantitative and qualitative questions about their child's experience and differences seen in the aquatic group

SECONDARY OUTCOMES:
Sensory Processing Measure (SPM: Preschool version: SPM-P, newer edition: SPM-2) Assessment Scores | Parents completed SPM on their child before the 8-week group began.
  Assessment given to parents to fill out before their child could start the aquatic group. Gives information on different sensory systems. Categories are: vision, hearing, touch, taste and smell, body awareness, balance and motion, sensory total, planning and ideas, and social participation. Interpretive range is: Typical, Moderate difficulties, and Severe difficulties.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen M Pataki, OTD, Principal Investigator — Cleveland State University
Locations (1):
- Seven Hills Recreation Center, Seven Hills, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
Not sure if other researchers will want access to this data.